CLINICAL TRIAL: NCT03257215
Title: A Phase IV, Double-blind, Randomised, Placebo-controlled Trial to Assess the Efficacy and Safety of Stoss Versus Daily Dose Oral Vitamin D Compared to Placebo for the Treatment of Atopic Dermatitis in Pre-school Aged Children- a Pilot Study
Brief Title: Can Vitamin D Treatment Help Treat Moderate to Severe Atopic Dermatitis in Young Children? the D-Vex Pilot Study
Acronym: D-Vex
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruitment very slow & ongoing funding not obtained.
Sponsor: Murdoch Childrens Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HREC 36237
Record Dates: First submitted 2017-08-13; First posted 2017-08-22 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Atopic Dermatitis
Keywords: Vitamin D
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Stoss vitamin D (Active Comparator): Stoss vitamin D at Day 1 and daily placebo for 90 days (Day 1 to 90)
  Interventions: Drug: Stoss vitamin D; Drug: Daily placebo
- Daily vitamin D (Active Comparator): Stoss placebo at Day 1 and daily vitamin D for 90 days (Day 1 to 90)
  Interventions: Drug: Daily vitamin D; Drug: Stoss placebo
- Placebo (Placebo Comparator): Stoss placebo at Day 1 and daily placebo for 90 days (Day 1 to 90)
  Interventions: Drug: Stoss placebo; Drug: Daily placebo

INTERVENTIONS:
Drug: Stoss vitamin D — A single 1.5 mL dose containing 150,000 IU cholecalciferol (100,000 IU/mL) administered on Day 1 (Solution in Olive Oil B.P. )
  Other Names: Stoss cholecalciferol
  Arms: Stoss vitamin D
Drug: Daily vitamin D — Daily 0.2 mL dose containing 1000 IU cholecalciferol administered from Day 1 to 90
  Other Names: Daily cholecalciferol (OsteVit D Liquid®)
  Arms: Daily vitamin D
Drug: Stoss placebo — A single 1.5 mL dose administered on Day 1
  Other Names: Oral Stoss Placebo (Olive Oil B.P.)
  Arms: Daily vitamin D; Placebo
Drug: Daily placebo — A once daily 0.2 mL dose administered from Day 1 to 90
  Other Names: Oral Daily Placebo (to match OsteVit D Liquid®)
  Arms: Placebo; Stoss vitamin D

SUMMARY:
Vitamin D is known to have a regulatory influence on both the immune system and skin barrier function. Studies in paediatric populations have found an inverse association of vitamin D levels and with both prevalence and severity of atopic dermatitis (AD). Trials of vitamin D as a treatment for AD are limited in number and size. There has never been a placebo-controlled randomised controlled trial of stoss high dose versus daily standard dose for the treatment of AD. Further, no trials have explored the presence of vitamin D pathway genes and response to treatment of AD. This pilot study will be used as a reference to determine outcomes and feasibility for undertaking a larger and more in depth definitive study.

ELIGIBILITY:
Inclusion Criteria:

* moderate to severe atopic dermatitis with a SCORAD ≥ 20 at baseline.
* aged between 1 ≤ 12 years of age at the time of randomisation.
* regularly ingest the recommended dietary intake (RDI) of calcium and plan to do so for the next 3 months
* have a legally acceptable representative capable of understanding the informed consent document and providing consent on the participant's behalf.

Exclusion Criteria:

* use of vitamin D supplementation, including a stoss dose of vitamin D in the previous year, or daily supplementation in the past month
* drink vitamin D fortified formula (all formulas) as the main milk intake
* received oral steroids within the past 6 months
* received oral immunosuppression in the past (cyclosporine, azathioprine, methotrexate)
* received UV therapy in the past 12 months
* have been fully formula fed within the past 6 months
* ave renal or liver or gastrointestinal (e.g.: coeliac, inflammatory bowel disease) disease
* receiving thiazide-type diuretics or anticonvulsant therapy
* have ever been diagnosed with Hypercalcaemia, Hypertension or Rickets
* unable to provide consent without the aid of an interpreter
* in the opinion of the Investigator, are unable to follow the protocol

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Change in SCORAD | Change from baseline at 3 months
  Atopic dermatitis severity score (SCORAD)

SECONDARY OUTCOMES:
Vitamin D levels | Baseline and 3 months
  vitamin D level in serum
Vitamin D polymorphisms | Baseline
  Presence of defined vitamin D polymorphisms
Immunoglobulin E (IgE) (serum) | Baseline and 3 months
  Serum
Effects on Parameters of bone metabolism (serum) | Baseline and 3 months
  Calcium, Phosphate, Parathyroid hormone, Alkaline Phosphatase
Effects on Parameters of bone metabolism (urine) | Baseline, 1 month and 3 months
  Calcium:Creatinine (urine)
Quality of life (family) | Baseline and 3 months
  Standardised questionnaire: Family Dermatology Life Quality Index (FDLQI)
Quality of life (child) | Baseline and 3 months
  Standardised questionnaire: Child Dermatology Life Quality Index (CDLQI) if >= 4 years of age OR Infant Dermatology Quality of Life (IDQOL) if <4 years of age
Compliance to study medications | Throughout the study period, , an average of 3 months
  Vitamin D stoss/daily and placebo stoss/daily
Adverse events | Throughout the study period, an average of 3 months
  Serious adverse events and serious adverse events
SCORAD | At 3 months
  Atopic dermatitis severity score (SCORAD)

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten P Perrett, MBBS, Principal Investigator — Murdoch Childrens Research Institute
Locations (1):
- Royal Children's Hospital Melbourne, Melbourne, Victoria, Australia